CLINICAL TRIAL: NCT04392583
Title: A Prospective, Multi-center, Single Arm Post-market Clinical Follow-up (PMCF) Study to Evaluate the Safety and Performance of ENTACT™ (Next Generation) Resorbable Septal Staple System for Septoplasty
Brief Title: Safety and Performance of ENTACT Septal Staple System for Septoplasty
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ENTACT.ENT.PRO.SEP.2019.05
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Septoplasty
Keywords: Septoplasty; ENTACT Septal Stapler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device: ENTACT Septal Staple: Septoplasty
  Interventions: Device: ENTACT Septal Staple system

INTERVENTIONS:
Device: ENTACT Septal Staple system — The ENTACT Septal Stapler delivers implantable septal staples which are intended to connect internal tissues to aid healing and for approximation of soft tissue during nasal septal surgery.

SUMMARY:
This is a prospective, multi-center, single arm PMCF study to evaluate the safety and performance of the ENTACT (Next Generation) resorbable staple system for septoplasty in 40 subjects. The study purpose is to provide evidence to satisfy the PMCF requirements of CE Marking to market this device in Europe (data may be used to support registrations on other countries as well).

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate clinical success of the ENTACT (Next Generation) resorbable septal staple system by examining the patient's nasal cavity at the 21 day follow-up visit.

The secondary objectives are to generate performance and health economics data to support the use of ENTACT (Next Generation) resorbable septal staple.

ELIGIBILITY:
Inclusion Criteria:

The patient will be eligible for the study if he or she meets all of the following inclusion criteria at the baseline screening:

1. Able and willing to give informed consent by voluntarily providing written informed consent in accordance with governing Institutional Review Board (IRB);
2. Clinically significant deviation of the nasal septum;
3. Willing and able to make all required study visits;
4. Able to read and understand the approved informed consent form and patient reported outcome assessments (written and oral)

Exclusion Criteria:

The patient will be ineligible for the study if he or she meets any of the following exclusion criteria at the baseline screening or during surgery:

1. Prolonged tissue approximation beyond that needed for normal tissue closure is necessary or desired;
2. Traditional suturing techniques are necessary;
3. Radiopacity is necessary or desired since ENTACT septal staples are radiotransparent;
4. Known to be allergic to foreign body of materials of investigational product;
5. Concomitant procedures other than turbinectomy, turbinate reduction, and/or sinus surgery;
6. Pregnancy at time of procedure;
7. Presence of infection at the site;
8. Severe drug and alcohol abusers;
9. Autoimmune disease deemed clinically significant by Principal Investigator (PI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population needing septoplasty
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharron E McCulloch, MS, Study Director — Smith & Nephew, Inc.; Stephan Mangin, Study Chair — Smith & Nephew, Inc.
Locations (3):
- United States (3):
  - ENT and Allergy Associates of Florida, Boca Raton, Florida
  - South Florida Sinus and Allergy Center, Fort Lauderdale, Florida
  - Beacon Medical Group Specialist, Elkhart, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sowerby LJ, Wright ED. A comparison of septal stapler to suture closure in septoplasty: a prospective, randomized trial evaluating the effect on operative time. Int Forum Allergy Rhinol. 2013 Nov;3(11):911-4. doi: 10.1002/alr.21209. Epub 2013 Aug 26. PMID 24039176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment for this study was conducted between 22 October 2020 and 25 June 2021 across three investigative sites.
Period: Overall Study
Arm/Group | Device: ENTACT Septal Staple
Started | 40
Completed | 39
Not Completed | 1
Not completed — Participant declined follow-up and subsequently withdrawn | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study (i.e., received the study device).
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (18.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Asian Indian | 0
  Race: Chinese | 0
  Race: Japanese | 0
  Race: Korean | 0
  Race: Southeast Asian | 0
  Race: Singaporean | 0
  Race: Indonesian | 0
  Race: Thai | 0
  Race: Cambodian | 0
  Race: Laotian | 0
  Race: Malaysian | 0
  Race: Filipino | 0
  Race: Vietnamese | 0
  Race: Myanmarese | 0
  Race: Bruneian | 0
  Race: Timor Lestian | 0
  Race: Other Asian | 0
  Race: Black or African American | 1
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: White | 37
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Success of the ENTACT Septal Staple System by Examining the Participant's Nasal Cavity at the 21 Day Follow-up Visit
Description: At the 21-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed YES or NO:
  * Septum wall straight appearance (yes/no)
  * Complete coaptation of perichondrial flaps on septum wall (yes/no)
  * Absence of significant local tissue reaction at the staple site (yes/no)
  * Absence of hematoma swelling at the staple site (yes/no)
  * No need for re-intervention at the surgery site (yes/no)
  If all the answers to the questions above were "YES" then clinical success was inferred (if any answer was "NO" then repair failure was inferred).
Time Frame: 21 days
Population: The Full Analysis Set (FAS) included participants enrolled in the study that had at least one post-baseline visit and were able to provide available data at the time frame specified.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 38
percentage of participants | 94.7 [82 to 99]

2. Secondary Outcome: Number of Participants With Septum Wall Straight Appearance at 5, 21, and 42-day Follow-up Visit (YES/NO)
Description: At the 5, 21, and 42-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed "YES" or "NO": Septum wall straight appearance.
Time Frame: Day: 5, 21, and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
Participants
  Day 5: number analyzed (Participants) | 37
  Day 5: Yes | 34
  Day 5: No | 3
  Day 21: number analyzed (Participants) | 38
  Day 21: Yes | 36
  Day 21: No | 2
  Day 42: Yes | 38
  Day 42: No | 1

3. Secondary Outcome: Number of Participants With Complete Coaptation of Perichondrial Flaps on Septum Wall at 5, 21, and 42-day Follow-up Visit (YES/NO)
Description: At the 5, 21, and 42-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed "YES" or "NO": Complete coaptation of perichondrial flaps on septum wall.
Time Frame: Day: 5, 21, and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
Participants
  Day 5: number analyzed (Participants) | 37
  Day 5: Yes | 35
  Day 5: No | 2
  Day 21: number analyzed (Participants) | 38
  Day 21: Yes | 38
  Day 21: No | 0
  Day 42: Yes | 39
  Day 42: No | 0

4. Secondary Outcome: Number of Participants With Absence of Significant Local Tissue Reaction at the Staple Site at 5, 21, and 42-day Follow-up Visit (YES/NO)
Description: At the 5, 21, and 42-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed "YES" or "NO": Absence of significant local tissue reaction at the staple site.
Time Frame: Day: 5, 21, and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
Participants
  Day 5: number analyzed (Participants) | 37
  Day 5: Yes | 35
  Day 5: No | 2
  Day 21: number analyzed (Participants) | 38
  Day 21: Yes | 38
  Day 21: No | 0
  Day 42: Yes | 39
  Day 42: No | 0

5. Secondary Outcome: Number of Participants With Absence of Hematoma Swelling at the Staple Site at 5, 21, and 42-day Follow-up Visit (YES/NO)
Description: At the 5, 21, and 42-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed "YES" or "NO": Absence of hematoma swelling at the staple site.
Time Frame: Day: 5, 21, and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
Participants
  Day 5: number analyzed (Participants) | 37
  Day 5: Yes | 37
  Day 5: No | 0
  Day 21: number analyzed (Participants) | 38
  Day 21: Yes | 38
  Day 21: No | 0
  Day 42: Yes | 39
  Day 42: No | 0

6. Secondary Outcome: Number of Participants With No Need for Re-intervention at the Surgery Site at 5, 21, and 42-day Follow-up Visit (YES/NO)
Description: At the 5, 21, and 42-day follow-up visit, the clinician examined the participant's nasal cavity and confirmed "YES" or "NO": No need for re-intervention at the surgery site.
Time Frame: Day: 5, 21, and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
Participants
  Day 5: number analyzed (Participants) | 37
  Day 5: Yes | 37
  Day 5: No | 0
  Day 21: number analyzed (Participants) | 38
  Day 21: Yes | 38
  Day 21: No | 0
  Day 42: Yes | 38
  Day 42: No | 1

7. Secondary Outcome: Nasal Obstructions Symptom Evaluation (NOSE) Score Collected at Pre-op and All Post-operative Visits
Description: The Nasal Obstruction Symptom Evaluation (NOSE) scale is a patient reported outcome (PRO). The NOSE Scale allows participants to quantify their symptoms based on the severity of their nasal obstruction/congestion. The NOSE score range was 0-100 were 0 represented no obstruction (i.e., better outcome) and 100 represented extreme obstruction (i.e., worse outcome).
Time Frame: Day: 0 (Screening), 5, 21 and 42
Population: The Full Analysis Set (FAS) included participants enrolled in the study that had at least one post-baseline visit and were able to provide available data at the time frame specified. Last Observation Carried Forward (LOCF) method was only used to carry forward post-baseline data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
score on a scale
  Screening | 69.2 (20.28)
  Day 5 | 62.5 (23.33)
  Day 21 | 39.9 (19.13)
  Day 42 | 33.2 (20.56)

8. Secondary Outcome: Visual Analog Scale (VAS) Pain Score Collected at Pre-Op and All Post-Operative Visits
Description: The Visual Analog Scale (VAS) for pain is a continuous scale completed by the participant who is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Scores range from 0-100 where a score of 0 represented no pain and a score of 100 indicated the worst pain possible.
Time Frame: Day: 0 (Screening), 5, 21 and 42
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
score on a scale
  Screening | 9.6 (19.82)
  Day 5 | 13.9 (20.92)
  Day 21 | 6.0 (12.40)
  Day 42 | 2.0 (5.78)

9. Secondary Outcome: Total Operation Time for the Procedure Overall and by Surgery Procedure Combinations
Description: Intra-operative surgery duration overall and by each surgery procedure combination (Septoplasty with Turbinate Reduction and Sinus Surgery, Septoplasty with Turbinate Reduction, Septoplasty with Sinus Surgery and Turbinectomy, and Septoplasty Alone) were recorded as time in minutes between start of the procedure and when the drapes are removed from the patient.
Time Frame: During procedure, up to 97 minutes
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
minutes
  Overall | 43.7 (27.88)
  Septoplasty with Turbinate Reduction and Sinus Surgery: number analyzed (Participants) | 18
  Septoplasty with Turbinate Reduction and Sinus Surgery | 64.9 (23.23)
  Septoplasty with Turbinate Reduction: number analyzed (Participants) | 16
  Septoplasty with Turbinate Reduction | 20.4 (7.31)
  Septoplasty with Sinus Surgery and Turbinectomy: number analyzed (Participants) | 2
  Septoplasty with Sinus Surgery and Turbinectomy | 67.0 (12.73)
  Septoplasty alone: number analyzed (Participants) | 3
  Septoplasty alone | 25.0 (15.72)

10. Secondary Outcome: Operative Closure Time With ENTACT Septal Stapler Procedure Overall and by Surgery Procedure Combinations
Description: Intra-operative time to deploy staples overall and by each surgery procedure combination (Septoplasty with Turbinate Reduction and Sinus Surgery, Septoplasty with Turbinate Reduction, Septoplasty with Sinus Surgery and Turbinectomy, and Septoplasty Alone) were recorded as time in seconds between start of closure to when the stapler was handed back to the scrub nurse.
Time Frame: During procedure, up to 306 seconds
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Device: ENTACT Septal Staple
Number analyzed (Participants) | 39
seconds
  Overall | 57.6 (54.81)
  Septoplasty with Turbinate Reduction and Sinus Surgery: number analyzed (Participants) | 18
  Septoplasty with Turbinate Reduction and Sinus Surgery | 82.2 (65.86)
  Septoplasty with Turbinate Reduction: number analyzed (Participants) | 16
  Septoplasty with Turbinate Reduction | 28.1 (12.06)
  Septoplasty with Sinus Surgery and Turbinectomy: number analyzed (Participants) | 2
  Septoplasty with Sinus Surgery and Turbinectomy | 125.0 (22.63)
  Septoplasty alone: number analyzed (Participants) | 3
  Septoplasty alone | 22.0 (4.58)

ADVERSE EVENTS:
Time Frame: Time of surgery (i.e. when device used) through end of the study (6 week post-operative follow-up).
Description: The Safety population (SAF) was used to analyze adverse events and included all enrolled participants who received the study device.
Arm/Group | Device: ENTACT Septal Staple
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: ENTACT Septal Staple (N=40)
PURULENT DRAINAGE OVER LEFT ANTERIOR ETHMOID (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device
COVID-19 (General disorders) | 1 (1) — Unrelated to device
COUGH (General disorders) | 1 (1) — Unrelated to device
FATIGUE (General disorders) | 1 (1) — Unrelated to device
RIGHT NASAL SCAR BAND (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device
EPISTAXIS (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device

LIMITATIONS AND CAVEATS:
No limitations reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT04392583/Prot_SAP_000.pdf